CLINICAL TRIAL: NCT04920773
Title: Community-based Post-exposure Prophylaxis for COVID-19: Results and Implications of Ayurveda Practice Guidelines
Brief Title: Community-based Post-exposure Prophylaxis for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Aarogyam UK (Other); Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University (Other); Samta Ayurveda Prakoshtha, India (Unknown); Padmanabhama Ayurveda Hospital and Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMP/CARE/01
Record Dates: First submitted 2021-06-06; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Post Exposure Prophylaxis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ayurveda Care Group (Experimental): Practice guidelines to follow physical distancing, respiratory and hand hygiene, wear mask Samshamani vati or Giloy Ghanavati
  Interventions: Other: Guduchi Ghanvati; Other: Standard guidelines
- Usual Care Group (Active Comparator): Practice guidelines to follow physical distancing, respiratory and hand hygiene, wear mask
  Interventions: Other: Standard guidelines

INTERVENTIONS:
Other: Guduchi Ghanvati — 500 mg of Samshamani vati or Giloy Ghanavati (Aqueous extract of Tinospora cordifolia) twice daily
  Arms: Ayurveda Care Group
Other: Standard guidelines — Practice guidelines to follow physical distancing, respiratory and hand hygiene, wear mask

SUMMARY:
Specifically identified Ayurvedic preparations is recommended by ministry of AYUSH as post-exposure prophylaxis to efficaciously prevent a negative person who has come into contact with COVID-19-positive. Traditionally, recommended Ayurvedic preparations have been used as antioxidants, antimicrobial and anti-inflammatory properties. Particularly, Guduchi Ghanvati has been recognised with its ability to control viral attachment, viral replication and induce immune response in pre clinical settings, and found to be one among the most important drugs in Ayurveda to fight against COVID-19.

However, known gap in guideline implementation and its impact on preventing active infection in exposed cases is unclear. Study aimed to increase the use of recommended AYUSH guidelines by having registered AYUSH physicians provide these medications, when indicated, in community based participants after known exposure to the SARS-CoV-2 coronavirus.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 60 years of age
* Household contact residing with the index case in the 14 days prior to index diagnosis within a residence without maintaining social distance
* Access to device and internet for telephonic appointments and follow up

Exclusion Criteria:

* Currently hospitalised
* Symptomatic with fever, cough, or shortness of breath
* Use of anti-malarial treatment or chemoprophylaxis
* Moderately or Severely ill for any co-morbid condition requiring medical assistance.
* Cognitive impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-06-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with active COVID-19 | 14-days following exposure
  PCR- proven COVID-19

SECONDARY OUTCOMES:
Time to symptoms onset | 14-days
  Days until start of symptoms of COVID-19
Disease Severity | 14 days
  Visual Analog Scale of rating overall symptom severity (0 = no symptoms; 10 = most severe)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, Study Chair — Aarogyam UK; Skanthesh Lakshmanan, Study Chair — Niramaya clinic, India; Isha Goyal, Principal Investigator — NMP Medical Research Institute, India; Abijith Venu, Study Chair — Aarogyam UK; Sahil Singhal, Study Director — NMP Medical Research Institute; Abhimanyu Kumar, Study Director — Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University
Locations (2):
- India (2):
  - NMP Medical Research Institute, Jaipur, Rajasthan
  - Padmnabham Ayurveda Hospital & Research Center, Jaipur, Rajasthan